CLINICAL TRIAL: NCT03863340
Title: Trapezius Muscle Fatigue of Long Duration: a Likely Neuromuscular Control Issue
Brief Title: Short Interventions to Prevent Trapezius Muscle Fatigue in Computer Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Turin, Italy (Other); University of Lausanne (Other); University of Michigan (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 32003B_160207
Record Dates: First submitted 2018-12-14; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Muscle Fatigue; Trapezius Muscle Strain
Keywords: muscle fatigue; work-related disorders; trapezius myalgia; sustained working task; high-density EMG

STUDY DESIGN:
Intervention Model Description: Randomized controlled laboratory experiment. 30 subjects are randomly assigned to two full day experiments either starting with the conditions including additional short interventions or without them.
Masking Description: Participants were informed that the study investigates neuro-motor mechanisms but not about the more specific research questions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- short interruptions of work tasks (Experimental): randomly start with or without short interruptions on the first experimental day and without or with them on the second experimental day
  Interventions: Behavioral: interruptions of work tasks

INTERVENTIONS:
Behavioral: interruptions of work tasks — During each activity two interruptions/breaks were selected randomly from a set of ten predetermined actions:
  Active break types:
  * Move shoulder and upper back
  * Swing arms near the body
  * Three slow but forceful elevations of the shoulders, a relaxation exercise based on the principles developed by Jacobson
  * Stand up and stretch
  * Slowly turn head in all possible directions.
  Passive break types:
  * Tell a couple of jokes
  * Stand up and have a drink
  * Relaxing the trapezius
  * Questions on actual posture and feelings of comfort / discomfort.
  * A short rest on the couch

SUMMARY:
This study is expected to demonstrate that during experimental days of seated computer work sustained and focalized low-level muscle activity contributes to the development of long-lasting fatigue effects (and thus possible disorder). On days with and without frequent interruptions, signs of fatigue and the activity pattern of the trapeze muscle are registered and compared using electromyographic registrations of the trapezius muscle.

DETAILED DESCRIPTION:
30 healthy adults without chronic neck pain participated in a laboratory study designed to simulate two full workdays of computer work. Within each session, participants performed five 50-min working activities separated by 10-min breaks: i) Use a computer keyboard to type a text presented on the left side of the screen; ii) do the typing task with the desk height set10 cm above elbow height; iii) play the computer game Spider Solitaire implemented in Windows 10; iv) Stroop test (This test consists of reading the name of a color whose text is in a color different from the name. The color name was then selected from a multiple-choice panel displaying color names; v) the same online puzzle game was presented to all participants. Assembling the puzzle was performed by drag and drop actions. The work periods were not disrupted (on the "control day") whereas two short interruptions of 5-min were introduced at 1/3 and 2/3 of each working period on the "intervention day". During these interruptions, participants were asked to perform "muscle disrupting/relaxing" activities. For each experimental session a 30-min lunch break took place between the third and the fourth work periods. The specific sequence of work activity type and disrupting/relaxing activities was randomized across participants; however, for each participant the order of work activities remained the same for the two experimental sessions (control and intervention days). The order of control and intervention days was also randomized between participants.

A set of six measures were performed at specific time intervals during each experiment: before the first work activity, before and after lunch, immediately and 1 hour after the fifth (last) work activity: i) upper trapezius activation, assessed through the temporal EMG profile recorded by a single bipolar signal; and ii) through the spatio-temporal distribution of EMG activity detected by a 2D array of electrodes (64 channels); iii) muscle fatigue, quantified by changes in electrically induced muscle twitch force signals, iv) isometric performance, v) dynamic performance; iii) cognitive and physical load and stress level. In addition, personality traits (anxiety level), perceived workload and musculoskeletal symptoms were evaluated as covariates.

ELIGIBILITY:
Inclusion Criteria:

* healthy experienced computer workers

Exclusion Criteria:

* chronic pain (more than 30 days within the last 12 months according to the Nordic Questionnaire (Kuorinka et al 1987);
* pathologies of the neck,
* prior and actual shoulder or neck pain caused by an accident,
* skin disease in the neck or shoulder area,
* BMI > 30,
* sleep disorders (e.g. apnea, restless legs syndrome),
* use of medications such as psychotropic drugs, muscle relaxants or analgesics within the last 3 days prior to the experiment,
* pregnancy.
* any shoulder/neck pain on the day before the experiment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2016-09-05 (Actual); Study Completion 2016-09-05 (Actual)

PRIMARY OUTCOMES:
EMG profile recorded by a single bipolar electrode: Rest-time | Continuously from the beginning to 370 min (end) of the simulated working activity of both the control and intervention day
  Rest-time (percentage of time below 5% of the standard activity level). The percentage of registration time without any rest time is called sustained low level muscle activity.
Spatio-temporal distribution of EMG activity: Area of muscle activity | Continuously from the beginning to 370 min (end) of the simulated working activity of both the control and intervention day
  The spatio-temporal distribution of EMG activity is detected by a 2D array of electrodes (64 channels) and the following outcomes are determined:
  Area of muscle active region (n. of channels)
Muscle fatigue: Change of muscle twitch | Change between 30 min before the beginning of the simulated working activity and 30 min after the end of the simulated working activity of both the control and intervention day
  3-D muscle twitch acceleration pattern measured at the acromion
Muscle fatigue: Change of dynamic force control accuracy | Change between 30 min before the beginning of the simulated working activity and 30 min after the end of the simulated working activity of both the control and intervention day
  Force control accuracy (mean squared error between the produced force (N) and the target force (N)) in an isometric dynamic tracking task

SECONDARY OUTCOMES:
EMG profile recorded by a single bipolar electrode: Static activity | Continuously from the beginning to 370 min (end) of the simulated working activity of both the control and intervention day
  p10 (level of the 10th percentile of the trapezius muscle activity) as an indicator of static activity primarily associated with continuous activity of the same pool of motor units.
Spatio-temporal distribution of EMG activity: Magnitude of activity | Continuously from the beginning to 370 min (end) of the simulated working activity of both the control and intervention day
  The spatio-temporal distribution of EMG activity is detected by a 2D array of electrodes (64 channels) and the following outcomes are determined:
  Magnitude of activity of muscle active regions (RMS sEMG).
Spatio-temporal distribution of EMG activity: Number of active epochs | Continuously from the beginning to 370 min (end) of the simulated working activity of both the control and intervention day
  The spatio-temporal distribution of EMG activity is detected by a 2D array of electrodes (64 channels) and the following outcomes are determined: Number of active epochs
Muscle fatigue: Change of static force control | Change between 30 min before the beginning of the simulated working activity and 30 min after the end of the simulated working activity of both the control and intervention day
  Force control accuracy (mean squared error between the produced force (N) and the target force (N)) in isometric isotonic low level contraction
Muscle fatigue: Change of force control in ramp contraction | Change between 30 min before the beginning of the simulated working activity and 30 min after the end of the simulated working activity of both the control and intervention day
  Force control accuracy (mean squared error between the produced force (N) and the target force (N)) in isometric ramp contraction.

OTHER OUTCOMES:
Localized musculoskeletal discomfort | At the start, and 70min, 130min, 190min, 310min, 370 min after the beginning of the simulated working activity of both the control and intervention day
  head-neck-shoulders-lower back-elbows-wrists-hip-upper legs-knees-ankles-feet-discomfort rated on 10 cm visual analog scales (adapted from Nordic questionnaire (Kuorinka et al 1987)
Visual and general fatigue | At the start, and 70min, 130min, 190min, 310min, 370 min after the beginning of the simulated working activity of both the control and intervention day
  10 cm visual analog scales
Effort | At the start, and 70min, 130min, 190min, 310min, 370 min after the beginning of the simulated working activity of both the control and intervention day
  6-20 Borg scale (6= no effort, 20=maximal possible effort)
EMG profile recorded by a single bipolar electrode: Dynamic activity | Continuously from the beginning to 370 min (end) of the simulated working activity of both the control and intervention day
  p90 (level of the 90th percentile of the trapezius muscle activity) as an indicator of dynamic activity which may promote variability in the recruitment of motor units
Spatio-temporal distribution of EMG activity: Centroid of active regions | Continuously from the beginning to 370 min (end) of the simulated working activity of both the control and intervention day
  The spatio-temporal distribution of EMG activity is detected by a 2D array of electrodes (64 channels) and the following outcomes are determined: Centroid of active regions

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Läubli, MD, Principal Investigator — Federal Institute of Technology Zurich

IPD SHARING:
Plan to Share IPD: No